CLINICAL TRIAL: NCT01780350
Title: Assessment of the Implementation of the ResQGARD® Impedance Threshold Device by the San Antonio Fire Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Circulatory Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-BAA-11-1
Record Dates: First submitted 2012-07-19; First posted 2013-01-31 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Acute Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ResQGARD ITD (Experimental): Subjects receive a ResQGARD ITD.
  Interventions: Device: ResQGARD ITD

INTERVENTIONS:
Device: ResQGARD ITD — Patients eligible for the device will receive the ResQGARD attached to a facemask or mouthpiece. The patient will use the device, provided it is tolerated, until their blood pressure is stabilized as determined by EMS personnel.

SUMMARY:
This study is attached to a comprehensive quality assurance/quality improvement (QA/QI) program conducted by the Office of the medical director, and is designed to contribute to generalizable knowledge to determine effectiveness and tolerability of an FDA approved Impedance Threshold Device (ITD) device in a large urban emergency medical service (EMS) system. The cohort will comprise a convenience sample of patients that are being treated by EMS for a hypotensive emergency.

ELIGIBILITY:
Inclusion Criteria:

* adults between the ages of 18-120 years
* presenting to EMS with or development of Hypotension during EMS interaction
* treated by EMS with the ITD

Exclusion Criteria:

* pediatric patients
* patients that do not present with or develop hypotension
* patients who the ITD will not form a secure seal due to anatomical abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ResQGARD ITD
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ResQGARD ITD
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 108
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline (Before ITD Use)
Description: Determining whether the application of an ITD will provide improvement in systolic blood pressure in subjects with hypotension in patients being treated by San Antonio EMS when compared to baseline.
Time Frame: During device use, up to 1 hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ResQGARD ITD
Number analyzed (Participants) | 200
mmHg | 17.9 (20.9)

2. Secondary Outcome: Tolerability
Description: Determine patient tolerability of the device while breathing through it. This is subjectively measured by the paramedic administering the device based on verbal reporting from the patient and paramedic estimation of the patient response to the device.
Time Frame: Duration of device use, up to 1 hour
Measure: Number; unit: participants
Arm/Group | ResQGARD ITD
Number analyzed (Participants) | 200
participants
  easy | 115
  moderate | 36
  difficult | 30
  not answered | 19

ADVERSE EVENTS:
Arm/Group | ResQGARD ITD
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No